CLINICAL TRIAL: NCT07391540
Title: Ekorostudien - Internet-based Cognitive Behavioral Therapy for Psychological Symptoms Related to Economy
Brief Title: ICBT for Psychological Symptoms Related to Economy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ekorostudien
Record Dates: First submitted 2026-01-13; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Depression and Anxiety Symptom
Keywords: Internet-based cognitive behavioral therapy (ICBT); Psychological treatment; Economy; Depression
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: All included participants will undergo the treatment simultaneously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): All included participants will undergo eight weeks of ICBT with weekly support by a therapist.
  Interventions: Behavioral: Internet-based cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioral therapy — The treatment consists of eight treatment modules that the participants receive, one module each week in eight weeks. The modules consists of texts, pictures and interactive exercises. The participants also get weekly guidance by a therapist and they can contact their therapist during the week if needed.
  Other Names: ICBT

SUMMARY:
This study aims to investigate the effects of guided internet-based cogitive behavioral therapy (ICBT) on psychological symptoms related to economy. In this pilot study, the investigators investigate participants' psychological symptoms before and after, and one and two years after, they have received eight weeks of therapist guided ICBT.

DETAILED DESCRIPTION:
The treatment the investigators investigate has been developed from earlier treatments used in studies that have shown to be effective for symptoms of depression, anxiety, and stress, among others. Participants will in this pilot study undergo ICBT with weekly guidance by a therapist and in a within-group design, the investigators will compare their self-reported psychological symptoms from before and after the treatment. A one- and two-year follow-up are also planned.

ELIGIBILITY:
Inclusion Criteria:

* Experience mild to moderate psychological symptoms or problems related to economy
* 18 years or older
* Ability to speak, read and write in Swedish
* Have access to the internet and a smartphone, computer or other device

Exclusion Criteria:

* Severe psychiatric or somatic illness that makes participation harder or impossible
* Ongoing addiction
* Acute suicidality
* Other ongoing psychological treatment
* Recent (within the latest month) changes in the dose of psychotropic medication or planned change of dose during the treatment weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
InCharge Financial Distress/Financial Well-Being Scale | Participants will complete this questionnaire at baseline, immediately after treatment, one year after treatment, and two years after treatment completion.
  The InCharge Financial Distress/Financial Well-Being Scale is a measure aiming to measure distress related to the individual's economic situation. It contains of eight questions where the respondent gets to answer on a scale from 1 to 10. This score is then divided by eight (number of questions) and total score is between 1 and 8. A higher score indicates better financial well-being.
Mongomery-Asberg Depression Rating Scale - Självrapportering | Participants will complete this questionnaire at baseline, immediately after treatment, one year after treatment, and two years after treatment completion.
  The Mongomery-Asberg Depression Rating Scale - Självrapportering is a self-report questionnaire that aim to measure symptoms of depression. It consists of 9 items and the repondent answers on a scale from 0 to 6. Scoring range is between 0-54. A higher score indicates more (severe) depression symptoms.
Generalized Anxiety Scale-7 item scale | Participants will complete this questionnaire at baseline, immediately after treatment, one year after treatment, and two years after treatment completion.
  The Generalized Anxiety Scale-7 item scale aim to measure anxiety symptoms and worry. When summing the points of the seven first questions, the scores are interpreted as mild, moderate and severe anxiety symptoms at 5-10, 11-15 and above 15 respectively. Thus, a higher score indicates higher levels of anxiety and worry. Total score range is between 0 and 21.

SECONDARY OUTCOMES:
Perceived Stress Scale-14 | Participants will complete this questionnaire at baseline, immediately after treatment, one year after treatment, and two years after treatment completion.
  The Perceived Stress Scale-14 is a questionnaire that aims to measure symptoms of stress. I contains 14 items that are scored on a range betewwn 0 (never) to 4 (very often). The total score range is between 0-56 and a higher score reflects higher levels of perceived stress.
Insomnia Severity Index | Participants will complete this questionnaire at baseline, immediately after treatment, one year after treatment, and two years after treatment completion.
  The Insomnia Severity Index is a measure of insomnia severity and symptoms of disordered sleep. Norm score ranges include low likelihood of sleep problems (0 to 7 points), some sleep problems (8 to 14 points), moderate sleep problems (15 to 21 points), and severe sleep problems (22 to 28 points). Thus, a higher score indicates more symptoms of insomnia. The score range is between 0 and 28.
Brunnsviken Brief Quality of Life Scale | Participants will complete this questionnaire at baseline, immediately after treatment, one year after treatment, and two years after treatment completion.
  The Brunnsviken Brief Quality of Life Scale is a measure of quality of life with a total score ranging from 0 to 96, with a higher score indicating a higher quality of life. The scores of each of the six primary questions regarding perceived quality of life within an area of life are multiplied by the score of an item measuring the perceived importance of the area in question.
Goldberg's (1999) International Personality Item Pool representation of Costa McCrae's (1992) Neuroticism-Extraversion-Openness Personality Inventory - Revised Domains | Participants will complete this questionnaire at baseline, immediately after treatment, one year after treatment, and two years after treatment completion.
  The Goldberg's (1999) International Personality Item Pool representation of Costa McCrae's (1992) Neuroticism-Extraversion-Openness Personality Inventory - Revised Domains is a measure of neuroticism. It consists of 10 items, scored from 0 (Very inaccurate) to 4 (Very accurate). A higher score indicates neurotic traits to a greater extent. The total score ranges from 0 to 40.
Rosenberg's Self-esteem Scale | Participants will complete this questionnaire at baseline, immediately after treatment, one year after treatment, and two years after treatment completion.
  The Rosenberg's Self-esteem Scale is a measure of self-esteem, consisting of ten items where five of them are positively and five of them are negatively worded. Sum scores range between 0 and 30. A higher score indicates higher self-esteem.

OTHER OUTCOMES:
Alcohol Use Disorder Identification Test | This measure was only used for screening purpose and was thus not included in the result analysis. Thus, it was only used at baseline.
  The Alcohol Use Disorder Identification Test is a 10-item screening tool to assess alcohol consumption, drinking behaviors, and alcohol-related problems. 10 items and scores ranging from 0-40, with higher scores indicating a higher level of alcohol use.
Knowledge test (created by the research team) | Participants will complete this questionnaire at baseline, immediately after treatment, one year after treatment, and two years after treatment completion.
  The knowledge test is a test about cognitive behavior therapy and how strategies in cognitive behavior therapy can be applied in everyday situations. It consists of 16 questions, and the respondent gets three answer options, with one of the alternatives being correct. The respondents also answer whether they are guessing/quite certain/entirely sure of their answer. The total score ranges between 0 and 16 for raw scores, and between -16 and 32 when certainty wheighted in.
Patient Health Questionnaire-4 | Used as a weekly measure of depression and anxiety during the treatment weeks. This questionnaire is only planned to be used for monitoring the participants' well-being, thus, it will not be included in the result analysis.
  The Patient Health Questionnaire-4 is a short self-report screening tool that consists of two questions about depressive symptoms and two questions about anxiety symptoms. It combines the first two questions in Patient Health Questionnaire-9 and the first two questions in the Generalized Anxiety Disorder-7 item scale. The items are answered on a scale from 0 to 3. Higher scores reflect more symptoms of depression and anxiety. Total score ranges between 0 and 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping, Östergötland County, Sweden